CLINICAL TRIAL: NCT01288183
Title: Behavioral Impact of Prefrontal Anodal Transcranial Direct Current Stimulation on Smokers
Brief Title: Anodal Transcranial Direct Current Stimulation (tDCS) in the Treatment of Tobacco Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Principal Investigator, Dr. E. Poulet, PUPH, Hôpital le Vinatier
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-A00180-39
Record Dates: First submitted 2011-01-27; First posted 2011-02-02 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Addiction; Smoking
Keywords: tobacco; smoking; tDCS; DLPFC
MeSH Terms: conditions — Behavior, Addictive; Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sham tDCS (Sham Comparator): sham transcranial direct current stimulation The anode (7 x 5 cm) is placed on the right dorsolateral prefrontal cortex. A large cathode (10 x 10cm) is placed on the left occipital region
  Interventions: Procedure: sham tDCS
- active tDCS (Active Comparator): active anodal tDCS over the right dorsolateral prefrontal cortex The anode (7 x 5 cm) is placed on the right dorsolateral prefrontal cortex. A large cathode (10 x 10cm) is placed on the left occipital region Intensity of the stimulation: 2 mA Duration of the stimulation: 20 min 10 sessions, 2 per day
  Interventions: Procedure: active tDCS

INTERVENTIONS:
Procedure: sham tDCS — sham condition as delivered by the stimulator "study mode" (2mA during 40s and brief current pulses until the end of the stimulation) 20 minutes, 10 sessions, 2 per day
  Arms: sham tDCS
Procedure: active tDCS — anodal tDCS applied over the right DLPFC 2mA, 20minutes, 10 sessions, 2 per day
  Arms: active tDCS

SUMMARY:
The aim of this study is to determine whether a powerful technique of noninvasive brain stimulation, transcranial direct current stimulation (tDCS), could reduce cigarette smoking and constitute a treatment of tobacco addiction.

DETAILED DESCRIPTION:
Tobacco is estimated to cause more than 5 millions yearly deaths in the developed world. Although most smokers would like to quit, relapse rates remain high. It seems that this relapse is linked with the process of craving, which is a powerful desire to smoke elicited by smoking deprivation or exposure to situations or cues that are associated with smoking. Neuroimaging studies have shown that the dorsolateral prefrontal cortex (DLPFC), and especially the right part, is critically involved in processing the craving of smoking. Increasing the activity of the DLPFC by noninvasive brain stimulation has been demonstrated to be effective in decreasing craving symptoms in cigarette smokers.

The aim of this study is to determine whether a powerful technique of noninvasive brain stimulation, transcranial direct current stimulation (tDCS), could reduce cigarette smoking. tDCS is a painless and safe brain stimulation method capable of modulating cortical excitability. The nature of these modulations depends on stimulation polarity: anodal tDCS is thought to cause neuronal depolarisation and thus enhancing cortical excitability whereas cathodal stimulation is proposed to reduce excitability. The investigators hypothesize that anodal tDCS applied repetitively to the right DLPFC could constitute a treatment of tobacco addiction. Therefore, the investigators will conduct a sham-tDCS-controlled, randomized, double-blind study.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 55 years old
* Tobacco consumption from 10 to 25 cigarettes, for at least 1 year
* Strong tobacco dependence at the Fagerstrom Test (score >= 5)
* Motivation to quit with a score >=12 at the Motivation to Quit Smoking Scale (Q-MAT)
* Informed consent

Exclusion Criteria:

* Concomitant Axe I psychiatric disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV)
* Other addictive disorder (DSM IV)
* No history of smoking cessation drug the previous year
* Psychotropic treatment
* Pregnancy or nursing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Smoking | Baseline (three days before starting tDCS regimen) to one-month after
  Self-reported number of cigarettes smoked each day

SECONDARY OUTCOMES:
Exhaled carbon monoxide | Baseline, one-week (after the last tDCS session) and one-month later
  measured using a CO monitor (MicroCo, Milford, MA, USA).
Craving | For each of the 10 tDCS sessions: Baseline and 0 hour post-tDCS (immediately after)
  measured using a 5-item Likert-type scale questionnaire of smoking urge
fMRI brain reactivity during a smoking cue-reactivity task | Baseline and one-week (after the last tDCS session)
  measured using an event-related fMRI paradigm

CONTACTS AND LOCATIONS:
Overall Officials: JEROME BRUNELIN, PhD, Study Director — Hopital le Vinatier; Emmanuel POULET, MD, PhD, Principal Investigator — Hopital le Vinatier
Locations (1):
- Hopital le Vinatier, Bron, France